CLINICAL TRIAL: NCT04751266
Title: Examination of Metal Contamination After Minimally Invasive Repair of Pectus Excavatum (MIRPE) and the Clinical Relevance
Brief Title: Metal Contamination After Minimally Invasive Repair of Pectus Excavatum (MIRPE)
Status: Completed | Type: Observational
Sponsor: Dr. Caroline Fortmann (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Sponsor-Investigator, Dr. Caroline Fortmann, Principal Investigator, Hannover Medical School
Organization: Hannover Medical School (Other)
Other Study IDs: 6659
Record Dates: First submitted 2016-01-13; First posted 2021-02-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Congenital Funnel Chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MIRPE: first minimally invasive repair of pectus excavatum
  Interventions: Procedure: minimally invasive repair of pectus excavatum

INTERVENTIONS:
Procedure: minimally invasive repair of pectus excavatum — substernal insertion of a metal bar

SUMMARY:
The purpose of this study is to determine whether there is a metal wear debris after minimally invasive repair of pectus excavatum and if there's a clinical relevance. Our hypothesis is that the metal bar after minimally invasive repair of pectus excavatum leads to a locally and systemic immune reaction due to elevated metal contamination.

ELIGIBILITY:
Inclusion Criteria:

* MIRPE

Exclusion Criteria:

* none

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
change of mean chromium values in blood (µg/l) | 4 years
  measurement of:
  1) chromium in blood (in µg/l)
  at the time points:
  1. pre implantation
  2. 4 weeks after implantation (to see change to baseline)
  3. 1 year after implantation (to see change to baseline)
  4. 2 years after implantation (to see change to baseline)
  5. explantation (usually 3 years after implantation; to see change to baseline)
  6. 6-12 months after explantation (to see change to explantation)
  We will compare the mean metal values at each time point post implantation with the mean metal values pre implantation. Clinical data like body weight etc. won't be relevant for the analysis.
change of mean chromium values in urine (µg/l) | 4 years
  measurement of: 2) chromium in urine (in µg/l)
  at the time points:
  1. pre implantation
  2. 4 weeks after implantation (to see change to baseline)
  3. 1 year after implantation (to see change to baseline)
  4. 2 years after implantation (to see change to baseline)
  5. explantation (usually 3 years after implantation; to see change to baseline)
  6. 6-12 months after explantation (to see change to explantation)
  We will compare the mean metal values at each time point post implantation with the mean metal values pre implantation. Clinical data like body weight etc. won't be relevant for the analysis.
change of mean chromium values in tissue (µg/g) | 3 years
  measurement of: 3) chromium in tissue (in µg/g)
  at the time points:
  1. implantation
  2. explantation (usually 3 years after implantation; to see change to baseline)
  We will compare the mean metal values at explantation with the mean metal values before implantation. Clinical data like body weight etc. won't be relevant for the analysis.
change of mean nickel values in blood (µg/l) | 4 years
  measurement of: 4) nickel in blood (in µg/l)
  at the time points:
  1. pre implantation
  2. 4 weeks after implantation (to see change to baseline)
  3. 1 year after implantation (to see change to baseline)
  4. 2 years after implantation (to see change to baseline)
  5. explantation (usually 3 years after implantation; to see change to baseline)
  6. 6-12 months after explantation (to see change to explantation)
  We will compare the mean metal values at each time point post implantation with the mean metal values pre implantation. Clinical data like body weight etc. won't be relevant for the analysis.
change of mean nickel values in urine (µg/l) | 4 years
  measurement of: 5) nickel in urine (in µg/l)
  at the time points:
  1. pre implantation
  2. 4 weeks after implantation (to see change to baseline)
  3. 1 year after implantation (to see change to baseline)
  4. 2 years after implantation (to see change to baseline)
  5. explantation (usually 3 years after implantation; to see change to baseline)
  6. 6-12 months after explantation (to see change to explantation)
  We will compare the mean metal values at each time point post implantation with the mean metal values pre implantation. Clinical data like body weight etc. won't be relevant for the analysis.
change of mean nickel values in tissue (µg/g) | 3 years
  measurement of: 6) nickel in tissue (in µg/g)
  at the time points:
  1. implantation
  2. explantation (usually 3 years after implantation; to see change to baseline)
  We will compare the mean metal values at explantation with the mean metal values before implantation. Clinical data like body weight etc. won't be relevant for the analysis.

SECONDARY OUTCOMES:
Observation of clinical reactions in correlation with elevated metal values | 4 years
  observation (description) of clinical symptoms of a metal allergy like
  * local rash
  * lassitude
  * chest pain
  * tachycardia
  * Nausea
  * pleural effusion
  for the time the bar is in place (3 years) and the metal values are evaluated.
  -> Then compare the mean metal values (see above) with the baseline and the other patients (with and/or without problems)
  No records when the patients don't have any problems.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Fortmann, MD, Principal Investigator — Department of Pediatric Surgery